CLINICAL TRIAL: NCT03874754
Title: Assessment of a Tailored Home-Based Exercise Program on Symptoms, Well-Being, and Resilience Among Cancer Survivors With Multiple Chronic Conditions
Brief Title: Tailored Home-Based Exercise Program for Multiple Chronic Conditions
Acronym: iHBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: J1886; P30NR018093-01 (NIH); IRB00175781 (Other: JHM IRB)
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Hypertension; Diabetes
Keywords: Multiple chronic conditions
MeSH Terms: conditions — Neoplasms; Hypertension; Diabetes Mellitus; Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: This is a two-arm parallel assignment involving two groups of participants. One group receives exercise intervention, and the other group receives usual care (control group).
Who Masked: Outcomes Assessor
Masking Description: Single blinded marking: The data collectors are blinded to the group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The iHBE program group (Experimental): Tailored Technology-Enhance Home-based exercise program (iHBE)
  Interventions: Other: Tailored Technology-Enhance Home-based exercise program (iHBE)
- Usual Care (Control group) (No Intervention): Participants were required to wear physical activity tracker (Fitbit) and respond to the daily symptoms survey (mEMA) while receiving usual care

INTERVENTIONS:
Other: Tailored Technology-Enhance Home-based exercise program (iHBE) — The tailored technology enhanced home-based exercise (iHBE) program is a 12-week program with 1 assessment home visit session, 5 home visits and 7 phone follow ups during exercise. The technologies, a wearable device, and a smartphone application, will be used as a tool to monitor physical performance (heart rate [HR], step count), provide immediate feedback, send daily reminding message through Mobile Ecological Momentary Assessment (mEMA). The coded raw data without personal identification information from the wearable device will be sent to the servers where the investigators can store it in the database alongside the mEMA data and create custom reports showing Heart Rate (HR) 30 minute before each Ecological Momentary Assessment (EMA) survey, showing HR and previous self-report responses before/ after each automatically triggered EMA.
  Other Names: iHBE
  Arms: The iHBE program group

SUMMARY:
A home-based, tailored, technology-enhanced home-based exercise program (iHBE) using a combination of the integrated mobile technologies (wearable device and phone application) and tailored home-based exercise will be pilot tested. Participants will choose one of the four home-based exercise options [National Institute of Aging (NIA) Go4Life (an exercise and physical activity campaign from the NIA), Iyengar-style yoga, walking, and modified Otago exercise] based on participants' preference and goals. The integrated mobile technologies system will allow the investigators to extract heart rate data directly from the wearable device to the research server. This data will be used to provide appropriate and personalized feedback on physical performance. The survey and notification to the participants on the smartphone.

DETAILED DESCRIPTION:
The benefits of physical activity on managing chronic illnesses and multiple symptoms are well established. However, increasing the physical activity of persons living with Multiple Chronic Conditions (MCC), especially low -income cancer survivors with MCC, is challenging. Home-based exercise improves physical activity and symptoms among persons with the single chronic disease. One major challenge of the home-based exercise is the motivation and adherence. The mobile technologies (e.g., wearable device and smartphone application) have been used to improve motivation and monitor a person physical activity. Guided by the society to cells framework and previous preliminary findings, the investigators developed a technology-enhanced home-based exercise program using a combination of the integrated mobile technologies (wearable device and phone application) and tailored home-based exercise. Participants will choose one of the four home-based exercise options [National Institute of Aging (NIA) Go4Life, Iyengar-style yoga, walking, and modified Otago exercise] based on participants' preference and goals. The integrated mobile technologies system will allow the investigators to extract heart rate data directly from the wearable device to the research server. This data will be used to provide appropriate and personalized feedback on physical performance and trigger algorithms to send the survey and notification to the participants in real time. This pilot project will examine the feasibility of this technology-enhanced home exercise tailored to participants' goals and preferences. The intervention will leverage the cancer survivorship phase (post-treatment) to motivate self-care by combining tailored existing evidence-based physical activity programs and mobile technology for participants to engage in the resilience-enhancing physical activity. Identification of BDNF's role as one of the exercise outcomes provide a novel target for an intervention and increase the investigators' understanding of the underlying mechanism of symptoms and resilience. This study aims to examine the feasibility and acceptability of the iHBE program among low-income cancer survivors living with co-morbid conditions. Eight participants who have completed treatment for a solid tumor cancer with at least one comorbidity (e.g., diabetes and/or hypertension) will be assigned to an open-label trial of the idea. The investigators will gather feedback on goal setting, problem-solving strategies, exercise choices, and tracking mechanisms, program feasibility, and acceptability and modify the intervention as needed.

ELIGIBILITY:
Inclusion Criteria:

* participants diagnosed with solid tumor cancer who have completed cancer treatment at least 6 months;
* diagnosed with diabetes and/or hypertension for at least a year;
* aged 21 years or older,
* have an annual household incomes of below $50,000 for families of three,
* the average fatigue level within the past 7 days at the level of 3 or more on the 0 (no fatigue) to 10 (worse fatigue) Likert scale
* give informed consent.

Exclusion Criteria:

* currently undergoing treatment for cancer;
* have an active infection (e.g., fever, localized redness, swelling, sinus congestion);
* diagnosed with a psychological disorder (e.g., suicidal or homicidal tendencies, extreme anxiety or depression)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nada Lukkahatai, PhD, Principal Investigator — Johns Hopkins School of Nursing
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared with other researchers

RESULTS

PARTICIPANT FLOW:
Groups:
- The iHBE Program Group: Tailored Technology-Enhance Home-based exercise program (iHBE): The tailored technology-enhanced home-based exercise (iHBE) program is a 12-week program with 1 assessment home visit session, 2 home visits on the first and last week of the program and 10 weekly phone follow up. Participants were asked to choose their methods of exercise and set up weekly goals for exercise with the researcher. The technologies, a wearable device, and a smartphone application were used as a tool to monitor physical performance (heart rate [HR], step count), provide immediate feedback, and send daily reminding messages through Mobile Ecological Momentary Assessment (mEMA). The physical performance and goals were reviewed and adjusted by both participant and researcher weekly.
Period: Overall Study
Arm/Group | The iHBE Program Group | Usual Care (Control Group)
Started | 22 | 12
Completed | 14 | 6
Not Completed | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The iHBE Program Group | Usual Care (Control Group) | Total
Number analyzed (Participants) | 22 | 12 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 20 | 11 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.73 (7.69) | 74 (4.79) | 73.18 (6.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 20 | 12 | 32
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 7 | 19
  White | 9 | 5 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 12 | 34
Fatigue [Mean (Standard Deviation); unit: T-score] — Fatigue will be assessed using the PROMIS Short Form v1.0 - Fatigue 6a, a 6-item self-report instrument that measures fatigue frequency, duration, and intensity, as well as its impact on physical, mental, and social activities. Each item is rated on a 5-point Likert scale (1 = never to 5 = always). Raw scores are converted to standardized T-scores (mean = 50, standard deviation = 10) based on the U.S. general population, with higher scores indicating greater fatigue.
  T-score | 52.64 (9.89) | 45.17 (7.93) | 50.15 (9.81)
Resilience [Mean (Standard Deviation); unit: units on a scale] — Resilience was measured by the 10-item Connor-Davidson Resilience Scale (CD-RISC-10), a self-report measure with items rated from 0 ('not true at all') to 4 ('true nearly all the time'). The total score ranges from 0 to 40, with higher scores indicating greater resilience.
  units on a scale | 35.56 (7.32) | 38.11 (8.43) | 36.41 (7.64)
Physical well-being [Mean (Standard Deviation); unit: units on a scale] — Physical well-being was assessed using the SF-36 Health Survey. The physical component summary was scored from the domains of physical functioning, role limitations due to physical health, and bodily pain (each ranging from 0 to 100). The average score were use for physical health score, with higher scores indicating better physical health.
  units on a scale | 42.52 (28.20) | 54.37 (32.40) | 48.44 (30.09)
Mental well-being [Mean (Standard Deviation); unit: units on a scale] — Mental well-being was assessed using the SF-36 Health Survey. Scores from the domains of vitality, social functioning, role limitations due to emotional problems, and mental health (each ranging from 0 to 100) were averaged to create a composite mental well-being score, with higher scores indicating better mental health.
  units on a scale | 73.66 (16.25) | 54.15 (38.50) | 63.91 (30.37)

OUTCOME MEASURES:

1. Primary Outcome: Change in Fatigue as Assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0-Fatigue 6a
Description: Fatigue was assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0-Fatigue 6a. This 6-item measure covers fatigue frequency, duration, intensity, and impact on daily activities. Responses were summed to generate a raw score (range 6-30), which was converted to a standardized T-score (mean = 50, SD = 10) based on the U.S. general population. Higher T-scores indicate greater fatigue (worse outcome). The reported outcome is the change in PROMIS Fatigue T-score from baseline to completion, where negative values indicate improvement.
Time Frame: Pre- and post-intervention, up to 12 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | The iHBE Program Group | Usual Care (Control Group)
Number analyzed (Participants) | 22 | 12
T-score | -1.61 (6.75) | 4.26 (7.95)

2. Primary Outcome: Change in Resilience as Assessed by Connor-Davidson Resilience Scale
Description: Resilience was assessed using the Connor-Davidson Resilience Scale (CD-RISC; 10 items). Each item is rated on a 5-point Likert scale (0 = not true at all to 4 = true nearly all the time). Raw scores are summed to produce a total score ranging from 0 to 40, with higher scores indicating greater resilience (better outcome). The reported outcome is the mean change in raw score, calculated as the score at the completion time point (12 weeks) minus the score at baseline. Positive values indicate improvement in resilience.
Time Frame: Pre- and post-intervention, up to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The iHBE Program Group | Usual Care (Control Group)
Number analyzed (Participants) | 22 | 12
score on a scale | 0.00 (4.97) | 0.89 (6.41)

3. Primary Outcome: Change in Physical Well Being
Description: Physical well-being was assessed using the 36-Item Short Form Health Survey (SF-36). The measure was derived from the physical functioning, role-physical, and bodily pain domains. Each domain is scored from 0 to 100, with higher scores indicating better physical health. The reported outcome is the mean change in the averaged domain scores from baseline to completion. Positive values indicate improvement in physical well-being.
Time Frame: Pre- and post-intervention, up to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The iHBE Program Group | Usual Care (Control Group)
Number analyzed (Participants) | 22 | 12
score on a scale | 14.48 (26.48) | -2.83 (17.67)

4. Primary Outcome: Change in Mental Well Being
Description: Mental well-being was assessed using the 36-Item Short Form Health Survey (SF-36). The Mental Component Score was calculated as the average of relevant domains (vitality, social functioning, role limitations due to emotional health, and mental health). Each domain is scored from 0 to 100, and the average domain score was used to represent overall mental well-being. Higher scores indicate better mental health. The reported outcome is the mean change in the averaged raw score from baseline to completion. Positive values indicate an improvement in mental well-being.
Time Frame: Pre- and post-intervention, up to 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | The iHBE Program Group | Usual Care (Control Group)
Number analyzed (Participants) | 22 | 12
score on a scale | 2.51 (6.29) | 0.16 (16.21)

5. Secondary Outcome: Physical Activity
Description: The physical activity will be measured in a form of average step count/day measured by a wrist-worn wearable device.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | The iHBE Program Group | Usual Care (Control Group)
Number analyzed (Participants) | 22 | 12
steps/day | 1279.11 (2986.71) | 805.46 (1682.42)

6. Secondary Outcome: Change in Brain-Derived Neurotrophic Factor Level (in Serum)
Description: The level of Brain-Derived Neurotrophic Factor in serum was measured by ELISA. The level will be measured in nanograms/milliliter.
Time Frame: Pre-and post-intervention, up to 12 weeks
Population: Due to the pandemic interruption with in-person research activity, we were unable to collect blood and sweat samples from the participants. Therefore, no data is available for this outcome.
Arm/Group | The iHBE Program Group | Usual Care (Control Group)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Brain-Derived Neurotrophic Factor Level (in Sweat)
Description: Brain-Derived Neurotrophic Factor level in sweat collected through the sweat pad. The level will be measured in nanograms/milliliter.
Time Frame: Pre- and post-intervention, up to 12 weeks
Population: as for outcome 6
Arm/Group | The iHBE Program Group | Usual Care (Control Group)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected within 6 months from baseline study visit
Arm/Group | The iHBE Program Group | Usual Care (Control Group)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/12
Other Adverse Events (participants affected / at risk) | 0/22 | 0/12

LIMITATIONS AND CAVEATS:
The study was interrupted by the COVID-19 pandemic, which led to unanticipated pauses in study activities and affected participant enrollment, intervention delivery, and follow-up assessments. As a result, the sample size was smaller than originally planned and some study procedures were modified. These factors may limit the generalizability of the findings and the ability to fully determine the intervention's effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/54/NCT03874754/Prot_SAP_000.pdf